CLINICAL TRIAL: NCT01053247
Title: Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel Group Study of 0416 Ointment.
Brief Title: Study of 0416 Ointment in the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0416
Record Dates: First submitted 2009-12-09; First posted 2010-01-21 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (Experimental): Test product that contains the active pharmaceutical ingredient
  Interventions: Drug: 0416
- Reference (Active Comparator): Reference product that contains active pharmaceutical ingredient
  Interventions: Drug: tacrolimus ointment 0.1%
- Vehicle (Placebo Comparator): Placebo that contains no active pharmaceutical ingredient
  Interventions: Drug: Vehicle of 0416 test product

INTERVENTIONS:
Drug: 0416 — Topical 0416 test product applied twice daily for 2 weeks
  Arms: Test
Drug: Vehicle of 0416 test product — Vehicle of 0416 test product applied twice daily for 2 weeks
  Arms: Vehicle
Drug: tacrolimus ointment 0.1% — Reference Product for 0416 test product. Apply twice daily for 2 weeks.
  Arms: Reference

SUMMARY:
The aim of this trial is to assess the efficacy of 0416 Ointment in the Treatment of Atopic Dermatitis.

Treatment medication will be administered as follows: Apply a thin layer of ointment to affected skin areas twice daily and rub in gently and completely. Study medication will be applied twice a day, approximately 12 hours apart, for approximately 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Atopic Dermatitis
* Good health with the exception of Atopic Dermatitis
* Percent Body Surface Area minimum requirements

Exclusion Criteria:

* Subjects who are pregnant, nursing, or planning a pregnancy within the study participation period.
* Subjects who have any systemic or dermatological disorders with the exception of Atopic Dermatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela C Kaplan, Study Director — Fougera Pharmaceuticals Inc.
Locations (1):
- Fougera Pharmaceuticals Inc., Melville, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test: Test product that contains the active pharmaceutical ingredient
  Tacrolimus Ointment 0.1% test product applied twice daily for 2 weeks
- Reference: Reference product that contains active pharmaceutical ingredient
  Protopic Ointment 0.1%: Reference Product applied twice daily for 2 weeks.
- Vehicle: Placebo that contains no active pharmaceutical ingredient
  Vehicle of Tacrolimus Ointment 0.1% applied twice daily for 2 weeks
Period: Overall Study
Arm/Group | Test | Reference | Vehicle
Started | 269 | 260 | 264
Completed | 249 | 241 | 236
Not Completed | 20 | 19 | 28
Not completed — Withdrawal by Subject | 9 | 4 | 15
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 2
Not completed — Lost to Follow-up | 8 | 5 | 7
Not completed — Adverse Event | 0 | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference | Vehicle | Total
Number analyzed (Participants) | 269 | 260 | 264 | 793
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 43.0 (16.29) | 43.7 (16.74) | 43.3 (17.14) | 43.3 (16.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 158 | 161 | 467
  Male | 121 | 102 | 103 | 326
Region of Enrollment [Number; unit: participants]
  United States | 258 | 253 | 255 | 766
  Central America | 11 | 7 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Success Based on the Investigator's Global Evaluation at the End of Treatment
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Test | Reference | Vehicle
Number analyzed (Participants) | 210 | 211 | 195
participants | 104 | 121 | 67

2. Secondary Outcome: The Mean Change From Baseline in the Total Individual Clinical Signs and Symptoms Per Body Region, the Mean Change From Baseline in Pruritus and Mean Change From Baseline in the Percentage Total Body Surface Affected (%BSA).
Time Frame: 2 weeks

ADVERSE EVENTS:
Arm/Group | Test | Reference | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/269 | 0/260 | 0/264
Other Adverse Events (participants affected / at risk) | 6/269 | 15/260 | 8/264
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=269) | Reference (N=260) | Vehicle (N=264)
Application Site Irritation (General disorders) | 3 | 6 | 0
Application Site Pruritus (General disorders) | 2 | 8 | 4
Atopic Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other